CLINICAL TRIAL: NCT06176820
Title: Vaginal Hyaluronic Acid, Arginine and Liposome Gel Versus Vaginal Lubricant in Postmenopausal Women With Genitourinary Syndrome of Menopause: A Prospective Double-blind Randomized Trial
Brief Title: Vaginal Hyaluronic Acid, Arginine and Liposome Gel Versus Vaginal Lubricant in Postmenopausal Women With Genitourinary Syndrome of Menopause
Acronym: VHAL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sarawak General Hospital (Other)
Responsible Party: Principal Investigator, Jun Jiet Ng, Obstetrician and Gynecologist, Principal investigator, Sarawak General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VHAL 001; NMRR ID-23-03429-ZXV. (Registry Identifier: National Medical Research Register)
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Menopause Related Conditions; Atrophic Vaginitis; Genitourinary Syndrome of Menopause; Sexual Dysfunction
Keywords: Genitourinary Syndrome of Menopause; Hyaluronic acid; Arginine; Liposome; Vaginal lubricant; Sexual Dysfunction; Vaginal Maturation Index; Vaginal Health Index
MeSH Terms: conditions — Atrophic Vaginitis; Sexual Dysfunction, Physiological | interventions — Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): Arm 1 will apply 2.5 gram of VHAL gel intravaginally using vaginal applicator 2 times per week for 3 months
  Interventions: Drug: Vaginal Gel
- Arm 2 (Active Comparator): Arm 2 will apply 2.5 gram of vaginal lubricant intravaginally using vaginal applicator 2 times per week for 3 months
  Interventions: Drug: Vaginal lubricant

INTERVENTIONS:
Drug: Vaginal Gel — Arm 1 will apply 2.5 gram of VHAL gel intravaginally using vaginal applicator 2 times per week for 3 months
  Arms: Arm 1
Drug: Vaginal lubricant — Arm 2 will apply 2.5 gram of vaginal lubricant intravaginally using vaginal applicator 2 times per week for 3 months
  Arms: Arm 2

SUMMARY:
The goal of this interventional study is to compare the efficacy and safety of vaginal hyaluronic acid, arginine and liposome gel versus vaginal lubricant in the treatment of genitourinary syndrome of menopause in postmenopausal women. The main question it aims to answer is:

Is vaginal hyaluronic acid, arginine and liposome gel more effective than vaginal lubricant in the treatment of genitourinary syndrome of menopause in postmenopausal women

Participants will be randomized into 2 treatment groups: vaginal hyaluronic acid, arginine and liposome group and vaginal lubricant group.

Researchers will compare whether vaginal hyaluronic acid, arginine and liposome group has better improvement than vaginal lubricant group.

DETAILED DESCRIPTION:
Ethical conduct of the study

The study will be conducted in compliance with the protocol and clinical research center (CRC) standard operating procedures. These are designed to ensure adherence to the ethical principles that have their origin in the "World Medical Association Declaration of Helsinki" (see Appendix), "Malaysian Guidelines for Good Clinical Practice" and applicable regulatory Requirements.

Informed consent and subject information

Freely given informed consent will be obtained from every participant prior to participation in this study. The investigator will inform every participant in detail about the nature of the study, its purpose, the treatments and the random assignment to treatment groups, those aspects of the study that are experimental, the procedures involved including the reasonably expected benefits the expected duration and the approximate number of participants involved and the participant's responsibilities. Written consent will be obtained from each participant involved in the study by the investigators in Gynecology clinic, Department of Obstetric and Gynecology, Sarawak General Hospital. If the subject and his/her parent/guardian are unable to read, the investigator or designee must explain to the subject the content of the Patient Information Sheet and Consent Form point by point in the presence of an impartial witness. The witness should personally sign and date the consent form. The participant will be given the opportunity to ask questions and time for consideration. A copy of the Patient Information Sheet and signed Consent Form will be given to the participant . The original will be filed by the principal investigator in the Investigator's Study File.

Patient data protection

The investigator will assure that the subjects' anonymity will be maintained and that the confidentiality of records and documents that could identify subjects will be protected, respecting the privacy and confidentiality rules in accordance with applicable regulatory requirements.

* Participants will be identified only by their assigned identification number.
* Investigators group 1 who are not blinded will keep a patient identification list with complete identification information (name, address, contact number, IC) on each subject.
* Participant's written informed consent form, should be maintained by the investigator in strict confidence.
* Study documents, records, and data will be kept in a locked locker in the Gynecology clinic. Electronic data will be kept in computer room 4 of Gynecology clinic which is password protected. Only investigators of VHAL study have access to the password.

Participants withdrawal & drop-out

Participants are free to withdraw from the study at any time for any reason. Participants may also be withdrawn from the study at any time at the discretion of the investigator. It should be understood that an excessive rate of withdrawals may render the study difficult to be interpreted. Missing data on efficacy assessments may significantly affect the interpretation of the study results. Should a subject withdraw or is withdrawn, every effort must be made to complete and report the observations as thoroughly as possible.

Possible reasons for withdrawal:

* Adverse event(s)
* Abnormal smear
* Improvement of subject's condition such that he/she no longer requires study treatment
* Insufficient therapeutic effect
* Protocol violation
* Participant requires use of unacceptable concomitant medication
* Participant not compliant with protocol procedures
* Participant develops a condition during the study that violates the inclusion/exclusion criteria
* Lost to follow-up
* Administrative problems
* Death
* Any other reason, in the investigator's opinion, that would impede the participant's participation in the study

Procedures for handling withdrawal

Participants who withdraw or are withdrawn from the study will:

* Have the reason(s) for their withdrawal recorded
* Be asked about the presence of any AEs and if so should be followed up by regular scheduled visits, telephone contact, correspondence or home visits until satisfactory clinical resolution of AEs is achieved.
* Be seen by an investigator and all final assessments will be performed and recorded in the Termination page of CRF.
* Be encouraged to continue coming for regular visits and assessments
* Have at least one follow-up contact (scheduled visit or telephone contact) for safety evaluation during the 30 days following the last dose of study treatment.
* Have study treatment returned

Participant replacement policy

There will be no replacement for subjects who withdraw or drop out

Treatment allocation and randomization

Recruitment Women with GSM presented to gynecology clinic. Patient Information Sheet with essential information on the trial will be provided to all potential participants. The recruiter will also provide any other information sought, emphasize the voluntary nature of participation, reinforce the point that care will not be affected if trial participation is declined and that the participant may withdraw from the study at any time without having to provide a reason and their subsequent care will not be affected in anyway. Written consent will be obtained from all who agreed to participate. Relevant demographic, medical data and VHAL Study Questionnaire will be collected as per the CRF.

Randomization

Randomization will be generated by random sequence generator, provided by random.org to avoid bias, and labelled on an opaque envelope, which will be taken out from a designated box upon recruitment of the patient, which will determine which arm the patient belongs to. Subjects will be randomized into 2 arms:

* Arm 1 with 26 participants will be assigned to VHAL gel
* Arm 2 with 26 participants will be assigned to vaginal lubricant

Double Blinding Investigators will be divided into 2 groups. Investigator group 1 will not be blinded and will be in charge of packaging, labeling of the investigation product and emergency unblinding procedures. Investigator group 2 will be in charge of recruitment, interview, examination and performing vaginal smear of the subjects. Investigator group 2 and subjects will be blinded to the study medication during the trial. Participants will not be told their allocated arm and will be given 2 tubes of 30 gram vaginal gel which are wrapped with white sticker to apply vaginally 2 times per weeks for 3 months.

Blinding & emergency unblinding procedures

Investigator group 2 and subjects will be blinded to the study medication during the trial. In the event that an adverse event (AE) occurs for which knowledge of the identity of the test drug is necessary to manage the subject's condition, the sealed emergency code key for that subject may be broken and the test drug identified by investigator group 1 who will be accessible at all times by telephone. Should emergency unblinding be required, the investigator group 2 will call investigator group 1 who will break the emergency code key for that subject, identify the test drug and inform the investigator group 2. A detailed report with the date and reason for identifying the study drug will be prepared by investigator group 1 and attached to the case report form (CRF). This report must be signed by investigator group 1 and investigator group 2 . All unused sealed code keys will be accounted for at the end of the study.

Except in the case of emergency, the blinding will be maintained until all subjects have completed the treatment and the database has been cleaned and locked. Any broken code will be clearly justified and explained by a comment on the case report form, along with the date on which the code was broken.

Baseline assessment and laboratory tests

Women with GSM presented to Gynecology clinic. Patient Information Sheet with essential information on the trial will be provided to all potential participants. The recruiter will also provide any other information sought, emphasize the voluntary nature of participation, reinforce the point that care will not be affected if trial participation is declined and that the participant may withdraw from the study at any time without having to provide a reason and their subsequent care will not be affected in anyway. Written consent will be obtained from all who agreed to participate. Relevant demographic, medical data and VHAL Study Questionnaire will be collected as per the CRF. The following criteria will be assessed during study enrollment.

* Social demographics, weight and height
* Co-morbid factors
* Primary disease
* Drug history
* Social history
* Sexual history

Assessment of compliance

Accountability and subject compliance will be assessed by maintaining adequate "drug dispensing" and return forms. A follow-up phone call will be made by investigator group 2 to check on the subject's compliance to vaginal gel/ vaginal lubricant application and side effects at 6 weeks of treatment. Subjects will be required to return all unused study medication to the investigator.

Detecting and documenting AE

Information about all AEs, whether volunteered by the patient, discovered by investigator questioning or detected through physical examination, laboratory test or other means, will be recorded on the Adverse Event Page of the CRF and followed up as appropriate

Information about all SAE will be recorded on the Serious Adverse Event Page of the CRF. All events documented in the SAE Form will be reported within 24 hours to the Clinical Research Centre (CRC)/sponsor by fax (see below for contact person and fax no.). The investigator will not wait to receive additional information to fully document the SAE before notifying CRC. A fax SAE form detailing relevant aspects of the SAE in question should follow telephone report of SAE. The investigator will also comply with the applicable regulatory requirements related to the reporting of unexpected serious drug reactions to the regulatory authorities. Where applicable, information from relevant medical records and autopsy reports will be obtained.

Any death, if brought to the attention of the investigator within 6 months after cessation of study treatment, whether considered treatment-related or not, will be reported to CRC.

Study contact for reporting SAE:

Name: Ho Kit Voon Department: Obstetric and Gynecology Tel: 082-276666 Fax: 082-242751 E-mail: kitvoonho@moh.gov.my Mobile phone: 018-667 9612

Treatment and follow up of AE

In the event of adverse effect, subjects may contact investigator Ho Kit Voon and proceed to Emergency Department, Sarawak General Hospital for assessment and treatment. If the adverse event occurs after the immediate application of the vaginal gel or lubricant, vaginal wash with normal saline will be performed to wash out the investigator's product. Investigator will follow up subjects with AE until the event has resolved or until the condition has stabilized. Appropriate medical care will be arranged for the patient. Abnormal tests will be repeated until they return to baseline levels or an adequate explanation of the abnormality has been found. Any follow up information will be reported to CRC monitor as soon as it becomes available.

Safety update

Investigator will notify all AEs that are serious or unexpected and very likely, probably or possibly related to the investigational product. The investigator will retain such notice with the Investigator's Brochure and immediately submit a copy of this information to the IRB/IEC. The IRB/IEC will determine if the informed consent requires revision. The investigator will also comply with the IRB/IEC procedures for reporting any other safety information.

Data management

Data management will be conducted using appropriate database and validation programs using computer in room 4 of Gynecology clinic which is password protected. Accurate and reliable data collection will be assured by verification and cross-check of 100% of the CRFs against the investigator's records (source document verification). The data collected will be entered into a computer database and subject to quality assurance procedures. Data entry, data validation, clean file and database lock will be carried out by investigator Rebecca Anak Tuloi.

Statistical methods

Sample size and power considerations The sample size calculation is based on a power of 80% (β=0.2), alpha of 0.05, in detecting a difference in change from baseline score of 0.7 between two groups with an assumed standard deviation (SD) of 0.85 for the primary efficacy endpoints (change from baseline in a composite score of vaginal dryness, soreness, irritation and dyspareunia) that is for a continuous outcome and equal sample size in both groups, the calculated sample size for each arm is 24 patients. Allowing for 10% dropout, a final sample size of 52 subjects with 26 subjects per arm will be used. The sample size is calculated based on the previous study by Ekin, M et al. (12).

Randomization

Randomization will be generated by a random sequence generator, provided by random.org to avoid bias, and labeled on an opaque envelope, which will be taken out from a designated box in the Gynecology clinic upon recruitment of the patient, which will determine which arm the patient belongs to. Subjects will be randomized into 2 groups:

* Arm 1 with 26 participants will be assigned to VHAL gel
* Arm 2 with 26 participants will be assigned to vaginal lubricant

Analysis The data analysis will be done using the SPSS version 22 by qualified statistician. Descriptive data will be expressed as mean ± standard deviation. Paired t-test and Wilcoxon-signed rank test will be used to compare before and after treatment. The efficacy of both groups will be compared using unpaired t-test and Mann-Whitney test. The results will be given in 95% confidence interval and considered significant if P < 0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with GSM,
* Postmenopause at least 1 year
* 40 to 80 years old

Exclusion Criteria:

* Vaginal smear with atypical cell
* The use of hormonal treatment/vaginal treatment in the previous 6 months
* History of hormone-dependent tumor
* Uninvestigated genital bleeding
* Smoker
* Serious disease/ chronic condition that interferes with study compliance

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological female
Enrollment: 52 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
The change in VHI Questionnaire score | The change in VHI Questionnaire score is assessed at the baseline visit and at 12 weeks of vaginal gel/ vaginal lubricant application
  Postmenopausal women with symptoms of genitourinary syndrome of menopause (GSM) will be asked to complete a questionnaire reporting their symptoms (vaginal pain, dyspareunia, vaginal dryness, burning, itching, and dysuria), and mark the severity of their symptoms on a 0-3 visual analogue scale (VAS). A score of 0 indicates the absence of a symptom, 1- mild , 2- moderate, 3-severe symptoms. We use the VHAL study questionnaire which is a modification of the validated vulvovaginal symptom questionnaire (VSQ-21).
The change in Vaginal Health Index (VHI) | The change in Vaginal Health Index (VHI) is assessed at the baseline visit and at 12 weeks of vaginal gel/ vaginal lubricant application
  The clinical evaluation will be performed by gynecologist blinded to the specific study-related information. The clinical data gathered included components of the Vaginal Health Index (VHI) score: elasticity, fluid secretion, potential of hydrogen (pH), epithelial mucosa integrity and moisture components. Each component is scored on a scale of 1 (worst) to 5 (best). The total score is 25 and lower scores indicate more severe atrophy. VHI will be calculated at baseline and 3 months after treatment.
The change in Vaginal Maturation Index (VMI) | The change in Vaginal Maturation Index (VMI) is assessed at the baseline visit and at 12 weeks of vaginal gel/ vaginal lubricant application
  Vaginal smear will be obtained from the upper one-third of the vagina using a spatula and stained according to the Papanicolaou technique at baseline and 3 months after treatment. The cytology samples will be fixed using alcohol and evaluated by an independent, blinded, board-certified pathologist from Department of Pathology, Sarawak General Hospital. The Vaginal Maturation Index (VMI) is determined by calculating the percentage of superficial, intermediate and parabasal epithelial cells on the smear by using this formula [(1 ×%superficial) + (0.5 × %intermediate) + (0 × %parabasal)]. The vaginal smear will be destroyed 3 months after the completion of study and will not be used for future study.

SECONDARY OUTCOMES:
Side effects of VHAL gel and vaginal lubricant | The side effects are assessed at the baseline visit and at 12 weeks of vaginal gel/ vaginal lubricant application
  * Systemic reactions such as anaphylaxis, generalized itchiness, urticaria
  * Local reactions such as stinging, burning, irritation or redness at the application site

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Portman DJ, Gass ML; Vulvovaginal Atrophy Terminology Consensus Conference Panel. Genitourinary syndrome of menopause: new terminology for vulvovaginal atrophy from the International Society for the Study of Women's Sexual Health and The North American Menopause Society. Climacteric. 2014 Oct;17(5):557-63. doi: 10.3109/13697137.2014.946279. Epub 2014 Aug 25. PMID 25153131
- [Background] Moral E, Delgado JL, Carmona F, Caballero B, Guillan C, Gonzalez PM, Suarez-Almarza J, Velasco-Ortega S, Nieto C; as the writing group of the GENISSE study. Genitourinary syndrome of menopause. Prevalence and quality of life in Spanish postmenopausal women. The GENISSE study. Climacteric. 2018 Apr;21(2):167-173. doi: 10.1080/13697137.2017.1421921. Epub 2018 Feb 7. PMID 29411644
- [Background] Ismael NN. A study on the menopause in Malaysia. Maturitas. 1994 Oct;19(3):205-9. doi: 10.1016/0378-5122(94)90073-6. PMID 7799827
- [Background] Harten IA, Evanko SP, Choe CH, Lee EW, Patel BN, Bogdani M, Wight TN, Lee UJ. The extracellular matrix molecules versican and hyaluronan in urethral and vaginal tissues in stress urinary incontinence. Neurourol Urodyn. 2021 Mar;40(3):771-782. doi: 10.1002/nau.24635. Epub 2021 Mar 1. PMID 33645869
- [Background] Nappi RE, Martella S, Albani F, Cassani C, Martini E, Landoni F. Hyaluronic Acid: A Valid Therapeutic Option for Early Management of Genitourinary Syndrome of Menopause in Cancer Survivors? Healthcare (Basel). 2022 Aug 13;10(8):1528. doi: 10.3390/healthcare10081528. PMID 36011183
- [Background] Cieri-Hutcherson NE, Jaenecke A, Bahia A, Lucas D, Oluloro A, Stimmel L, Hutcherson TC. Systematic Review of l-Arginine for the Treatment of Hypoactive Sexual Desire Disorder and Related Conditions in Women. Pharmacy (Basel). 2021 Mar 27;9(2):71. doi: 10.3390/pharmacy9020071. PMID 33801678
- [Background] Liu P, Chen G, Zhang J. A Review of Liposomes as a Drug Delivery System: Current Status of Approved Products, Regulatory Environments, and Future Perspectives. Molecules. 2022 Feb 17;27(4):1372. doi: 10.3390/molecules27041372. PMID 35209162
- [Result] Abdridged Life Tables Malaysia 2019-2021. Department of Statistics Malaysia, Official Portal. 2021